CLINICAL TRIAL: NCT00688623
Title: A Single Arm, Multicenter Single Stage Phase II Trial of RAD001 as Monotherapy in the Treatment of Metastatic Non Syndromic Neuro-endocrine Tumors
Brief Title: RAMSETE: RAD001 in Advanced and Metastatic Silent Neuro-endocrine Tumors in Europe
Acronym: RAMSETE/CDE16
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001CDE16
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Advanced and Metastatic Silent Neuro-Endocrine Tumors; Carcinoma; Neuroendocrine; Non Functioning Neuroendocrine Tumors (NETs); Non Syndromic Neuroendocrine Tumors; Carcinoids; Non Functioning
Keywords: Neuroendocrine tumors; non functioning neuroendocrine tumors; Non syndromic neuroendocrine tumors; carcinoids; non-functioning carcinoids; adults; everolimus; NET; RAMSETE; CRAD001; non-functioning neuroendocrine tumors carcinoids
MeSH Terms: conditions — Carcinoma; Carcinoid Tumor; Neuroendocrine Tumors | interventions — Everolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Everolimus (Experimental): Everolimus
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus 5 mg tablets were supplied in blister packs

SUMMARY:
To evaluate the preliminary efficacy and safety of RAD001 as monotherapy for first-line treatment of patients with metastatic papillary carcinoma of the kidney.

ELIGIBILITY:
Inclusion criteria:

1. ≥ 18 years old
2. Patients with advanced (unresectable or metastatic) biopsy proven non-syndromic neuro-endocrine carcinoma, low or intermediate grade
3. Radiological documentation of disease progression within 12 months prior to study entry. If patients received anti-tumor therapy during the past 12 months, they must have radiological documentation of progressive disease (PD) while on or after receiving the therapy
4. Patients may have received previous treatments (chemotherapy, biotherapy, peptide-receptor radionuclide therapy); an overall maximum of 3 systemic treatment is allowed
5. Patients with at least one measurable lesion
6. Patients with an ECOG (Eastern Cooperative Oncology Group) Performance Status 0-2
7. Adequate bone marrow function
8. Adequate liver function
9. Adequate renal function
10. Adequate lipid profile

Exclusion criteria:

1. Patients with poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoid and small cell carcinoma
2. Patients with carcinoid with hormone related symptoms (diarrhea ≥ 4 stools per day and/or flushes)
3. Patients with Islet cell carcinomas or pancreatic NET
4. Patients who received prior therapy with Vascular Endothelial Growth Factor (VEGF) pathway inhibitor within 4 weeks prior to study entry
5. Patients who entered peptide receptor radionuclide therapy (PRRT) within 3 months prior to study entry
6. Patients who received CT, biotherapy or radiotherapy within 4 weeks prior to study entry
7. Patients who have previously received systemic (mammalian target of rapamycin) mTOR inhibitors
8. Patients with a known hypersensitivity to everolimus or other rapamycins or to its excipients
9. Patients with uncontrolled central nervous system (CNS) metastases
10. Patients receiving chronic systemic treatment with corticosteroids or another immunosuppressive agent
11. Patients with a known history of HIV seropositivity
12. Patients with autoimmune hepatitis
13. Patients with an active, bleeding diathesis
14. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
15. Patients who have a history of another primary malignancy and off treatment ≤ 3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of the uterine cervix
16. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods
17. Patients who are using other investigational agents or who had received investigational drugs ≤ 4 weeks prior to study treatment start
18. Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-06-24 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2016-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (33):
- France (4):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Munich
- Italy (10):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Viagrande, CT
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Perugia
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Viagrande
- Novartis Investigative Site, Rotterdam, Netherlands
- Poland (2):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Warsaw
- Spain (4):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Uppsala
- Sweden (2):
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Glasgow - Scotland
  - Novartis Investigative Site, Manchester

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eighty-two patients were screened and 73 were treated with study drug.
Groups:
- Everolimus: 10 mg/day dose of everolimus was given by continuous oral daily dosing of two 5 mg tablets
Period: Overall Study
Arm/Group | Everolimus
Started | 73 (Intent to treat (ITT))
Safety Analysis Set | 73 (received at least one dose of study drug and had at least one post-baseline safety assessment)
Per Protocol (PP) | 60 (no major protocol deviation and 50% of planned dose of 8 weeks or d/c due to disease progression)
Completed | 18
Not Completed | 55
Not completed — Adverse Event | 22
Not completed — abnormal lab value | 1
Not completed — Withdrawal by Subject | 4
Not completed — Death | 3
Not completed — disease progression | 23
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 71
  Other | 2
Tumor histology/cytology [Count of Participants; unit: Participants]
  Bronchial (thymic) carcinoid -typical | 9
  Bronchial (thymic) carcinoid -atypical | 12
  Neuroendocrine tumor | 16
  Neuroendocrine carcinoma | 36
Time since first diagnosis [Count of Participants; unit: Participants]
  < 1 year | 19
  1 year to < 3 years | 26
  3 years to < 6 years | 17
  6 years to < 10 years | 3
  ≥ 10 years | 6
  Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants' Best Overall Response Rate at 12 Months - Per Protocol Set (PP)
Description: Overall response rate (ORR) was based on RECIST central assessment and defined as the percentage of patients with best overall response (BOR) of a confirmed complete response (CR) or partial response (PR). The BOR was calculated on basis of the tumor of overall lesion response evaluated at each visit. To be assigned a status of PR or CR, changes in tumor measurements had to be confirmed by repeat assessments obtained within 4 weeks after the criteria for response were first met. Assessments was based on RECIST criteria 1.0. Measurable disease lesions had to be accurately measured in at least one dimension with longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm with spiral CT scan (with minimum lesion size no less than double the slice thickness). PR required at least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters. CR required disappearance of all target and non-target lesions.
Time Frame: baseline up to approximately 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Everolimus
Number analyzed (Participants) | 60
percentage of participants
  Complete response (CR) | 0.0
  Partial response | 0.0
  Stable disease (SD) | 56.7
  Progressive disease (PD) | 43.3
  Unknown | 0.0

2. Primary Outcome: Percentage of Participants With Objective Response Rate at 12 Months - Per Protocol Set (PP)
Description: Overall Response Rate (ORR) was calculated for total PP population based on central review as confirmatory, primary analysis as well as for ITT population as sensitivity analysis. It was presented with relative frequencies and the exact 2-sided 80% confidence limit (CI) computed using the Clopper-Pearson method). If the lower limit of the CI did not include p0=5%, the hypothesis that p ≤ 5% was rejected. The primary analysis was based on the PP Set
Time Frame: baseline up to approximately 12 months
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Everolimus
Number analyzed (Participants) | 60
percentage of participants | 0.0 [0.0 to 3.8]

3. Primary Outcome: Percentage of Participants With a Overall Response Rate With a Complete Response (CR) or Partial Response (PR) at 12 Months ITT Set
Description: The best overall response (BOR) was calculated on basis of the tumor of overall lesion response evaluated at each visit. To be assigned a status of PR or CR, changes in tumor measurements had to be confirmed by repeat assessments that should have been performed not less than 4 weeks after the criteria for response were first met. Assessments was based on RECIST criteria 1.0. Measurable disease lesions had to be accurately measured in at least one dimension with longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm with spiral CT scan (with minimum lesion size no less than double the slice thickness). PR required at least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
  CR required disappearance of all target and non-target lesions.
Time Frame: baseline up to approximately 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Everolimus
Number analyzed (Participants) | 73
percentage of participants
  Complete response (CR) | 0.0
  Partial response | 0.0
  Stable disease (SD) | 74.0
  Progressive disease (PD) | 16.4
  Unknown | 9.6

4. Primary Outcome: Percentage of Participants With Objective Response Rate at 12 Months ITT Set
Description: Overall Response Rate (ORR) was presented for ITT population as sensitivity analysis. It was presented with relative frequencies and the exact 2-sided 80% confidence limit (CL; computed using the Clopper-Pearson method). If the lower limit of the CI did not include p0=5%, the hypothesis that p ≤ 5% was rejected.
Time Frame: baseline up to approximately 12 months
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Everolimus
Number analyzed (Participants) | 73
percentage of participants | 0.0 [0.0 to 3.1]

5. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR) at 12 Months for Per Protocol (PP) and ITT Sets
Description: DCR was based on central radiologic review and is defined as the percentage of patients with a best overall response of 'Complete response' (CR), 'Partial response' (PR) or 'Stable disease' (SD). Relative frequencies together with their exact 2-sided 80% confidence intervals were presented
Time Frame: baseline up to approximately 12 months
Population: subjects who met required criteria
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Everolimus
Number analyzed (Participants) | 73
percentage of participants
  DCR for Per protocol set: number analyzed (Participants) | 60
  DCR for Per protocol set | 56.7 [47.6 to 65.4]
  DCR for Intent to treat set | 50.7 [42.6 to 58.8]

6. Secondary Outcome: Percentage of Participants' Biochemical Response Rate Based on the Tumor Marker Chromogranin A (CgA)
Description: Biochemical response was defined as level and change from baseline in CgA during the course of the trial. The resulting values showed a high variation and were not interpretable, as different methodology was used for the assessment of CgA at the individual centers.
Time Frame: baseline up to approximately 12 months
Population: The resulting values showed a high variation and were not interpretable, as different methodology was used for the assessment of CgA at the individual centers.
Arm/Group | Everolimus
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Progression Free Survival (PFS) for Per Protocol (PP) and ITT Sets
Description: Duration of PFS was defined as the time from first study drug administration to objective tumor progression or death from any cause. Observations from patients not experiencing tumor progression or death at date of database closure were censored with the date of their last adequate tumor assessment. Progression was either 1) a 20% increase in the sum of the longest diameter of all target lesions, taking as reference the smallest sum of longest diameter of all target lesions recorded at or after baseline or 2) the appearance of a new lesion or 3) the unequivocal progression of non-target lesions.
Time Frame: baseline up to approximately 12 months
Population: subjects who met required criteria
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Everolimus
Number analyzed (Participants) | 73
days
  PFS days for Per protocol set: number analyzed (Participants) | 60
  PFS days for Per protocol set | 185 [160 to 262]
  PFS days for Intent to treat set | 190 [161 to 262]

8. Secondary Outcome: Overall Survival (OS) for Per Protocol (PP) and ITT Sets
Description: OS was defined as the time from first study drug administration to death from any cause. If a patient was not known to have died at date of database closure, overall survival was censored at the date of last contact.
Time Frame: baseline up to approximately 15 months
Population: subjects who met required criteria
Measure: Mean (Standard Error); unit: days
Arm/Group | Everolimus
Number analyzed (Participants) | 73
days
  OS for Per protocol set: number analyzed (Participants) | 60
  OS for Per protocol set | 451.8 (19.8)
  OS for Intent to treat set | 437.1 (18.6)

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse events are reported in this record from First Patient First Treatment until Last Patient Last Visit up to approximately 15 months
Arm/Group | Everolimus
Serious Adverse Events (participants affected / at risk) | 48/73
Other Adverse Events (participants affected / at risk) | 72/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=73)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphatic obstruction (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1
Retinal detachment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 5
Enteritis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 3
Intestinal perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 2
General physical health deterioration (General disorders) | 1
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden death (General disorders) | 1
Acute hepatic failure (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Febrile infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 2
H1N1 influenza (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pseudomonas infection (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Subdiaphragmatic abscess (Infections and infestations) | 1
Expired product administered (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Presyncope (Nervous system disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Astringent therapy (Surgical and medical procedures) | 1
Aortic rupture (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=73)
Anaemia (Blood and lymphatic system disorders) | 11
Tachycardia (Cardiac disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 18
Abdominal pain upper (Gastrointestinal disorders) | 9
Aphthous ulcer (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 30
Dry mouth (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 4
Mouth ulceration (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 22
Stomatitis (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 18
Asthenia (General disorders) | 19
Chest pain (General disorders) | 8
Chills (General disorders) | 5
Fatigue (General disorders) | 19
Mucosal inflammation (General disorders) | 18
Oedema (General disorders) | 5
Oedema peripheral (General disorders) | 15
Pain (General disorders) | 5
Pyrexia (General disorders) | 11
Conjunctivitis (Infections and infestations) | 4
Cystitis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 11
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 7
Blood glucose increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 5
Blood potassium decreased (Investigations) | 5
Blood thyroid stimulating hormone decreased (Investigations) | 5
Blood triglycerides increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 8
Haemoglobin decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 6
Weight decreased (Investigations) | 17
White blood cell count decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 23
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 12
Flank pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 10
Lethargy (Nervous system disorders) | 8
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 7
Onychoclasis (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 32
Flushing (Vascular disorders) | 4
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.